CLINICAL TRIAL: NCT03145077
Title: Using Magnetic Resonance Imaging (MRI) to Assess Mandibular and Soft Tissue Responses to Radiation Therapy
Brief Title: Dynamic Contrast-Enhanced Magnetic Resonance Imaging in Diagnosing Osteoradionecrosis in Patients With Head and Neck Cancer That Is Primary, Has Come Back, or Has Spread to Other Places in the Body
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PA16-0302; NCI-2018-02608 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA16-0302 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Osteoradionecrosis; ORN; Dynamic contrast-enhanced magnetic resonance imaging; DCE-MRI; Questionnaires; Surveys
MeSH Terms: conditions — Head and Neck Neoplasms; Osteoradionecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (DCE-MRI) (Experimental): Patients with newly diagnosed tumors undergo DCE-MRI within 4 weeks prior to the first radiation fraction, within 3-5 weeks after radiation start, and at 2, 6, 12, 24, and 36 months post radiation. Patients who were previously irradiated and are at various stages of oncologic follow-up undergo DCE-MRI for a total of 2-5 times at baseline and at 6, 12, 24, 36, and/or 48 months post radiation. Patients in the third or subsequent years post treatment may undergo subsequent yearly imaging studies.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Questionnaire Administration
- Cohort 2 (DCE-MRI) (Experimental): Patients undergo DCE-MRI within 4 weeks prior to the first re-radiation fraction, within 3-5 weeks after radiation start, and at 2, 6, 12, 24, and 36 months post radiation.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Questionnaire Administration
- Cohort 3 (DCE-MRI) (Experimental): Patients undergo DCE-MRI before and at 2 and 6 months post ORN treatment. Patients may undergo DCE-MRI during the mid-ORN treatment.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Questionnaire Administration
- Cohort 4 (DCE-MRI) (Experimental): Patients undergo DCE-MRI within 4 weeks prior to and at 5-10 weeks and 12 months post surgery.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE-MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) works in diagnosing osteoradionecrosis in patients with head and neck cancer that is primary, has come back, or has spread to other places in the body who are undergoing radiation therapy. DCE-MRI may help doctors to predict osteoradionecrosis in patient with head and neck cancer undergoing radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether DCE-MRI following external beam radiation therapy (EBRT) can be used to reliably predict osteoradionecrosis (ORN).

SECONDARY OBJECTIVES:

I. Define dose-response relationships between DCE-MRI derived imaging biomarkers and subsequent development of ORN.

II. Evaluate the use of DCE-MRI parameters to monitor ORN response to treatment.

III. Assess the use of DCE-MRI parameters in preoperative planning in advanced ORN subjects.

IV. Develop MRI-based biomarkers inclusive predictive models for development of radiotherapy-attributable tissue injury within the field of radiation.

V. Determine the association of patient-related outcomes (PROs) to clinical and imaging findings of tissue damage, such as the onset of ORN.

OUTLINE: Patients are assigned to 1 of 4 cohorts.

COHORT 1: Patients with newly diagnosed tumors undergo DCE-MRI within 4 weeks prior to the first radiation fraction, within 3-5 weeks after radiation start, and at 2, 6, 12, 24, and 36 months post radiation. Patients who were previously irradiated and are at various stages of oncologic follow-up undergo DCE-MRI for a total of 2-5 times at baseline and at 6, 12, 24, 36, and/or 48 months post radiation. Patients in the third or subsequent years post treatment may undergo subsequent yearly imaging studies.

COHORT 2: Patients undergo DCE-MRI within 4 weeks prior to the first re-radiation fraction, within 3-5 weeks after radiation start, and at 2, 6, 12, 24, and 36 months post radiation.

COHORT 3: Patients undergo DCE-MRI before and at 2 and 6 months post ORN treatment. Patients may undergo DCE-MRI during the mid-ORN treatment.

COHORT 4: Patients undergo DCE-MRI within 4 weeks prior to and at 5-10 weeks and 12 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Patients must have histologic evidence of malignant neoplasm that may have been obtained from the primary tumor or metastatic lymph node
* Receipt of external beam radiation therapy (EBRT) with curative intent, with or without concomitant chemotherapy
* Good performance status (Eastern Cooperative Oncology Group [ECOG] score 0-2)
* Willing to comply with all study procedures; and
* Willing to participate for the duration of the study
* COHORT 1 (LONGITUDINAL) GROUP 1 (PRE-RADIATION): Subjects who are currently undergoing or scheduled to undergo treatment with radiotherapy with or without chemotherapy (induction or concurrent) with intent to eradicate the malignancy. Treatment will include the following: 1) primary or nodal disease adjacent to (within 2 cm) the mandible (i.e., likely to receive a dose of at least 50 Gy to some portion of the mandible volumes) and 2) > 60% probability of survival for 3 years after treatment
* COHORT 1 (LONGITUDINAL) GROUP 2 (POST-RADIATION): Subjects who were previously treated with radiotherapy with or without chemotherapy (induction or concurrent). Treatment will have included the following: 1) unilateral maximum mandible dose of >= 60 Gy and a gradient of dose across the mandible of >= 20 Gy, 2) oncological cure and now in disease surveillance; and 3) no clinically diagnosed ORN at the time of enrollment
* COHORT 2 (ENRICHED): Subjects with recurrent and/or new head and neck cancer disease who will undergo re-irradiation to the head and neck with intent to eradicate the malignancy. Treatment will include the following: 1) any mandible dose of at least 50 Gy cumulative (initial and subsequent treatment); and 2) no clinically diagnosed ORN at the time of enrollment
* COHORT 3 (EARLY ORN INTERVENTION): Subjects with clinically confirmed low-grade/early stage osteoradionecrosis requiring therapeutic (medical and/or dental surgery) intervention as diagnosed by a qualified clinician. Clinical staging of developing or existing ORN will be conducted using the CTCAE 4.0 (Common Terminology Criteria for Adverse Events)
* COHORT 4 (SURGICAL INTERVENTION FOR ADVANCED ORN): Subjects with clinically confirmed high grade/high stage osteoradionecrosis requiring surgical intervention. Clinical staging of ORN will be conducted using the CTCAE 4.0 (Common Terminology Criteria for Adverse Events)

Exclusion Criteria:

* Unable to tolerate diffusion weighted (DW)-MRI or DCE-MRI
* Having an estimated glomerular filtration rate (GFR) < 60 ml/min/1.73 m^2
* Contraindication to MRI (e.g. non-MRI compatible metallic implants)
* Pregnant females and cognitively impaired patients
* Unable or unwilling to give written, informed consent to undergo MRI imaging
* Claustrophobia
* Unable to obtain imaging studies of adequate quality to assess imaging-based biomarkers
* COHORT 1/GROUP 1: Previously treated with radiotherapy for a malignant neoplasm of the head and neck, excluding cutaneous lesions. Determination will be made by review of the radiation therapy plan and dosimetry map to evaluate mandible exposure to radiation
* COHORT 1/GROUP 2: Previously treated with radiotherapy for a malignant neoplasm of the head and neck more than one time, excluding cutaneous lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
DCE-MRI Derived Parameters Following External Beam Radiation Therapy (EBRT) and Subsequent Development of Osteoradionecrosis (ORN) | 5 years
  Spatiotemporal parameter maps extracted from patient DCE-MRI scans.
  Clinical staging of developing or existing ORN conducted according to the CTCAE 4.0.

SECONDARY OUTCOMES:
Dose-Response Relationships Between DCE-MRI Derived Imaging Biomarkers and Subsequent Development of Osteoradionecrosis (ORN) | 5 years
  Voxel-by-voxel correlation of delivered radiation dose to mandible and DCE-MRI parameter changes determined to establish a dose-biomarker response relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lai, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Moreno A, Sahli AJ, Johnson F, Sun X, Barbon C, Rinsurongkawong W, Song W, Luciani FM, Liang H, Li J, Liu W, Lee JJ, Frank SJ, Lai S, Fuller C, Hutcheson K; P01 MD Anderson Oropharynx Cancer Program. Stiefel MD Anderson OroPharynx cancer (MDA-OPC) cohort: a single-institution, prospective longitudinal outcomes study. BMJ Open. 2025 Nov 24;15(11):e106845. doi: 10.1136/bmjopen-2025-106845. PMID 41290309
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org